CLINICAL TRIAL: NCT04919187
Title: Accuracy and rEliabilitY of the vEstibuLo-ocular ExAmination Performed by inteRNs IN the emerGency Department
Acronym: EYE LEARNING
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: EYE LEARNING
Record Dates: First submitted 2021-04-30; First posted 2021-06-09 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Acute Vestibular Syndrome; Emergencies
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Dizziness, loss of balance, and unsteadiness of gait are common symptoms reported by Emergency Department (ED) patients. The incidence of acute vestibular syndrome (AVS) is increasing and reaches 2-4% of ED visits. In the ED of the Paris Saint Joseph Hospital Group, its incidence was 5% during the year 2019 and 2% during the year 2020 (COVID-19 pandemic period).

Emergency medicine is based on a dichotomous principle for any acute pathology in the initial phase. For AVS, the diagnostic dilemma for emergency physicians is usually to differentiate a benign vestibular cause from a potentially serious cerebral cause such as ischemic stroke of the vertebro-basilar territory. The majority of AVS are related to acute vestibulopathies, yet it is necessary to recognize and distinguish a benign paroxysmal positional vertigo (BPPV) from a vestibular neuritis, a vestibular migraine, or a labyrinthine hydrops, to exclude with certainty a cerebral involvement. However, posterior fossa strokes mimic 5% of BPPV and 25% of vestibular neuritis. Among these strokes, about 20% are therefore revealed by a VAS without associated localizing neurological sign. In the absence of a clear neurological sign, the emergency physician must therefore decide whether to treat the patient as an outpatient when he or she suspects a AVS of "peripheral" origin (otolaryngology), or as an inpatient when he or she suspects a "central" origin, in particular a stroke.

DETAILED DESCRIPTION:
Unfortunately, the diagnostic evaluation of an isolated AVS is often frustrating because patients with vertigo tend to be uncertain and imprecise when describing their symptoms. Examination of the vestibulo-ocular pathway, by assessing eye movements in different head positions, is an essential step in the clinical examination to reliably and quickly predict the origin of a AVS. The 3-step clinical rule "HINTS" (Head Impulse, Nystagmus, Test of Skew) was developed in 2009 by "neuro-ophthalmologists" in the USA. It evaluates the vestibulo-ocular reflex by the Head Impulse Test (pathological with the presence of ocular saccades for a peripheral AVS), the characteristics of the nystagmus (multidirectional and/or vertical for a central AVS), and looks for ocular misalignment (Test of Skew with cover-test, pathognomonic of a central involvement). In patients at high cardiovascular risk, HINTS is 100% sensitive and 96% specific in predicting posterior fossa stroke within 2 minutes at the bedside, compared with the Gold-Standard. The "STANDING" (SponTAneous, Nystagmus, Direction, head Impulse test, STANDING) clinical rule is a structured bedside diagnostic algorithm in four clinical steps. It is based on the evaluation of two eye movements (Head Impulse Test and nystagmus), an evaluation of gait (search for ataxia) and the search for positional nystagmus (Dix Hallpike test for the posterior canal and Panigni test or "supine and roll test" for the lateral canal). In the ED, with patients at heterogeneous cardiovascular risk, the STANDING is more interesting than the HINTS. Indeed, it allows the detection of BPPV in pauci-symptomatic patients at the time of their clinical evaluation (i.e., those without spontaneous nystagmus). It had also shown excellent performance (sensitivity:95%, specificity:87-96%) in diagnosing any central cause of VAS in the hands of emergency physicians. However, the 2017 validation study of STANDING had an audit bias. The gold standard test, brain imaging, had only been performed when deemed appropriate (ie, in 34% of peripheral diagnoses, and for only 5% of these by brain MRI).

In the EYE-ECG study conducted at the GhPSJ SU from October 2019 to January 2021, the invesitgators determined the diagnostic performance of these two clinical rules performed by emergency physicians to 300 patients with isolated VAS, comparing it to the Gold-Standard. The manuscript of this study has been published in the Academic Emergency Medicine journal (DOI: 10.1111/acem.14337) in June 2021. Its originality was to evaluate the performance of the tests in the hands of emergency physicians and on a population not selected for its risk of stroke. The investigators showed that the HINTS and STANDING tests had excellent sensitivities (97% and 94% respectively) and negative predictive values (99% and 98% respectively) for predicting any central cause of VAS on brain MRI. They thus allowed emergency physicians to exclude a central cause in a rapid manner (on average 5±3 minutes) with very acceptable false-negative rates (3% and 6%, respectively), and with a potential impact on the reduction of unnecessary brain imaging (-33% and -32%, respectively). For predicting MRI normality, STANDING was more specific than HINTS (75% vs. 67%). This is explained by the addition of a clinical item dedicated to positional nystagmus in the STANDING, and by the high prevalence of BPPV among VAS of ENT origin in SU patients (40%). Indeed, among the false-positives of the HINTS test (erroneously predicted as a central cause for benign vestibular disease), one third of the diagnoses were BPPVs.

The major limitation of the EYE-ECG study was that it did not assess interindividual variability of the HINTS and STANDING tests between different emergency physicians. The STANDING validation study was the only study that assessed global and individual agreement of the algorithm item scores in a binary "central or peripheral" mode between two senior emergency physicians. The inter-observer agreement of the STANDING was good globally (K=0.83) and also at each step of the algorithm (distinction between spontaneous and positional nystagmus: K=0.83, interpretation of a multidirectional or vertical nystagmus: K=0.95, normal Head Impulse Test: K=0.74, recognition of a walking ataxia: K=0.81)18.

Each semester, an average of 7 medical students in general medicine and one in emergency medicine complete an internship at the GhPSJ. In routine practice, the medical students interview and examine their patients alone. They document their clinical examination in the patient's medical record and then present the patient's clinical record to a senior emergency physician. In a second step, the patient is clinically reassessed by the senior emergency physician who becomes responsible for the patient's diagnostic and therapeutic strategy. The accuracy of the vestibulo-ocular examination performed by medical students has never been described in the literature.

The hypothesis of the investigators is that after standardized theoretical training and with the clinical experience gained during their semester in the ED, medical students should be able to examine and interpret the vestibulo-ocular examination of patients with isolated AVS as accurately as seniors.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age is ≥ 18 years
* French-speaking patient.
* Patient presenting on admission to the emergency department with an isolated AVS defined by a course of more than one hour and less than one week and the presence of at least one symptom among:

  1. vertigo: an illusion of displacement of the subject in relation to surrounding objects or surrounding objects in relation to the subject, a sensation of rotation, displacement of the body in the vertical plane, instability described as pitching or as a "spinning head", sometimes associated with vegetative signs (nausea, vomiting, pallor, sweating, slowing of the heart rate)
  2. and/or spontaneous or positional nystagmus,
  3. and/or a gait disorder: such as imbalance with lurching, or a shaky gait, or simple instability.
* A patient may be included several times during the study period provided that they are distinct acute episodes of isolated AVS.

Exclusion Criteria:

* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection
* Patient objecting to the use of his/her data for this research
* Patient with focal neurological signs concomitant with AVS: a language or writing disorder, a speech disorder such as dysarthria, a disorder in the execution of voluntary movements, a sensory, motor or visual deficit, involuntary abnormal movements
* Patient with a history of oculomotor paralysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective diagnostic monocentric cohort study. These patients consulted the SU for symptoms integrated in an isolated AVS, i.e.: vertigo, balance disorder, instability on walking, present for at least one hour and less than one week, as defined by the Barany Society. The study will be reported using the STARD Statement criteria.
Sampling Method: Non-Probability Sample
Enrollment: 321 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-09-21 (Actual)

PRIMARY OUTCOMES:
To determine the diagnostic accuracy of the STANDING algorithm performed by ED medical student to distinguish central from peripheral causes of isolated AVS in the ED. | Day 1
  Sensitivity and specificity of the STANDING algorithm performed by ED medical student.

SECONDARY OUTCOMES:
To determine the inter-rater reliability of each items of the STANDING algorithm, between an ED medical student and a senior emergency physician for each patient. | Day 1
  Inter-observer agreement measured by the overall Fleiss Kappa coefficient (K) and by the K each item of the STANDING algorithm performed by the ED medical student and by the senior emergency physician
To evaluate the changing opinions of ED medical students on vestibulo-ocular examination between the beginning and the end of their internship in the ED | Day 1
  Changing confidences of the ED medical students regarding each item of the STANDING algorithm measured on a survey with a 5-points Likert scale, at the beginning and at the end of their ED internship

CONTACTS AND LOCATIONS:
Overall Officials: Camille GERLIER, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

REFERENCES:
- [Result] Gerlier C, Fels A, Vitaux H, Mousset C, Perugini A, Chatellier G, Ganansia O. Effectiveness and reliability of the four-step STANDING algorithm performed by interns and senior emergency physicians for predicting central causes of vertigo. Acad Emerg Med. 2023 May;30(5):487-500. doi: 10.1111/acem.14659. Epub 2023 Jan 30. PMID 36628557